CLINICAL TRIAL: NCT03519672
Title: Prospective Psychometric Evaluation Study of a Patient-reported Outcomes (PRO) Instrument for Congenital Thrombotic Thrombocytopenic Purpura (cTTP, Upshaw-Schulman Syndrome [USS], Hereditary Thrombotic Thrombocytopenic Purpura [hTTP]
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 281701
Record Dates: First submitted 2018-04-23; First posted 2018-05-09 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Congenital Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with cTTP - adolescents: Adolescents aged 12 to 17 years
  Interventions: Other: No intervention
- Participants with cTTP - adults: Adults aged ≥18 years
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The purpose of this study is to assess the psychometric properties of a recently developed congenital thrombotic thrombocytopenic purpura (cTTP)-specific patient-reported outcomes (PRO) instrument.

ELIGIBILITY:
Inclusion criteria:

1. The participant is an adolescent aged 12 to 17 years or an adult aged ≥18 years;
2. The participant has been diagnosed with congenital thrombotic thrombocytopenic purpura (cTTP) and is currently receiving prophylactic or on-demand treatment with fresh frozen plasma (FFP), or solvent detergent (S/D) plasma, or Von Willebrand Factor/Factor VIII (VWF/FVIII) concentrates;
3. In the instance that the participant is identified and recruited remotely (Direct-to-Patient (DtP) recruitment), access to the internet and possession of an internet-connecting device is required;
4. The participant has provided informed consent, and in the instance that the participant is an adolescent, a legal guardian has provided informed consent and the adolescent has provided assent.

Exclusion criteria:

1. The participant cannot read nor write;
2. The participant is non-English speaking;
3. The participant is currently participating in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified for inclusion by the Investigator (physician) and, if interested to participate, they will be asked to provide informed consent (and assent for adolescents 12 to 17 years). The legally authorized representative (LAR) of participating cTTP adolescents (ages 12 to 17 years) will provide informed consent on the adolescent's behalf. A qualified vendor will also be used to identify potentially eligible participants through various networks.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Quality of life (QoL) outcomes: cTTP-specific PRO instrument | Day 1, and Day 14
  The congenital thrombotic thrombocytopenic purpura (cTTP)-specific patient-reported outcomes (PRO) instrument consists of 26 questions designed to assess the patient's experience of fatigue, joint, muscle, abdominal and chest pain in the previous 24 hours, neurologic manifestations, bruising, feelings of depression and mood alterations, and activity limitation in the past 7 days, and patient's attitudes, experienced side effects, work/school absences and travel impact associated with treatment received for TTP during the previous 2 weeks.
Change from baseline of Quality of life (QoL) outcomes: PROMIS®-29 | Day 1, and Day 14
  The Patient-Reported Outcomes Measurement Information System (PROMIS®)-29 Profile is a collection of 4-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and the ability to participate in social roles and activities, as well as a single pain intensity item.
  The individual scales for fatigue, pain interference, anxiety and depression, each being 5-point Likert scales, and the single pain intensity item, a 0 to 10 Numerical Rating Scale, will be used in this study. A higher score for all these scales indicate poorer HRQL (worse symptoms).
Change from baseline of Quality of life (QoL) outcomes: Pediatric PROMIS® Subscales for adolescents | Day 1, and Day 14
  The Patient-Reported Outcomes Measurement Information System (PROMIS®)-29 Profile is a collection of 4-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and the ability to participate in social roles and activities, as well as a single pain intensity item. The Pediatric PROMIS® Subscales will be used for adolescents.
  The individual scales for fatigue, pain interference, anxiety and depression, each being 5-point Likert scales, and the single pain intensity item, a 0 to 10 Numerical Rating Scale, will be used in this study. A higher score for all these scales indicate poorer HRQL (worse symptoms).
Change from baseline of Quality of life (QoL) outcomes: HIT-6 | Day 1, and Day 14
  The Headache Impact Test (HIT)-6 is a short-form scale, partially derived from the 54-item HIT, and used to measure the impact of headaches in the past 4 weeks on the ability to function at work, at school, at home and in social situations. Items are scored on a 5-point Likert scale ranging from 6=Never, 8=Rarely, 10=Sometimes, 11=Very often, 13=Always, with a global score ranging from 36 to 78, a higher score indicating a worse HRQL.
Change from baseline of Quality of life (QoL) outcomes: Condensed MCMDM-1VWD Bleeding Questionnaire: Bruising Subscale | Day 1, and Day 14
  The Condensed MCMDM-1VWD Bleeding Questionnaire is a bleeding-specific questionnaire used to produce a bleeding score for von Willebrand disease, which was developed by eliminating all details not directly affecting the bleeding score from the validated and extensive MCMDM-1VWD questionnaire. This study will only use the 5 close-ended questions of the bruising scale. These 5 questions assess the presence of bruising (yes/no), location (exposed/unexposed sites) and average size (<1cm, 1 to 5cm and >5cm), presence of minimal or no trauma (yes/no), and whether medical attention was required (yes/no).
Change from baseline of Quality of life (QoL) outcomes: PDQ-5 | Day 1, and Day 14
  The Perceived Deficits Questionnaire 5-Item (PDQ-5) is a subscale of the full-length Perceived Deficits Questionnaire (PDQ), developed specifically for participants with Multiple Sclerosis to assess perceived cognitive deficits from the subject's perspective. The PDQ has 4 5-item subscales: Attention/Concentration, Retrospective Memory, Prospective Memory, and Planning/Organization. The PDQ-5 consists of the 5 PDQ items correlating most strongly with the total PDQ score; items from all 4 subscales are represented.
Change from baseline of Quality of life (QoL) outcomes: NEI-VFQ-25 | Day 1, and Day 14
  The National Eye Institute Visual Function Questionnaire (NEI-VFQ or VFQ)-25 is a valid and reliable 25-item version of the 51-item NEI-VFQ. The questionnaire measures the impact of visual impairment on Health Related Quality of Life (HRQL). The general vision (1 item), near vision (3 items), and distant vision activities (3 items) subscales will be used in this study. Each item is associated with a 6-point Likert scale ranging from 1 (no difficulty at all) to 6 (stopped doing this for other reason or not interested in doing this), and global scores range from 0 to 100, a higher score indicating better HRQL.
Change from baseline of Quality of life (QoL) outcomes: WPAI-GH | Day 1, and Day 14
  The self-administered Work Productivity and Activity Impairment-General Health (WPAI-GH) is a 6-item scale measuring work (5 items) and daily activities (1 item). Scores express the impairment percentage so a lower score represents more productivity.
Change from baseline of Quality of life (QoL) outcomes: WPAI-GH plus Classroom Impairment questions for adolescents | Day 1, and Day 14
  The Work Productivity and Activity Impairment (WPAI) plus Classroom Impairment Questionnaire will be used for adolescents. The WPAI plus Classroom Impairment Questionnaire measures school attendance; productivity levels at school; and ability to perform regular daily activities. The WPAI plus Classroom Impairment Questionnaire is a 9-item scale measuring school/work (8 items) and daily activities (1 item). Scores express the impairment percentage so a lower score represents more productivity. While the instructions from the instrument will not be changed, adolescent participants will be instructed to consider their school work and activities when completing the questionnaire.
Change from baseline of Quality of life (QoL) outcomes: PGI-S | Day 1, and Day 14
  The Patient Global Impression of Severity (PGI-S) is a 1-item questionnaire designed to assess participant's impression of disease severity that was adapted to congenital thrombotic thrombocytopenic purpura (cTTP). The PGI-S item asks the respondent to best describe how their cTTP symptoms severity is now Scores are on a 4-point scale scored as: "normal" (1), "mild" (2), "moderate" (3), or "severe" (4).
Change from baseline of Quality of life (QoL) outcomes: PGI-Change | Day 1, and Day 14
  The Patient Global Impression of Change (PGI-C) is a single 1 item questionnaire that compares the participant's current health state to when treatment was started. Response options range from 1 (Very Much Improved) through 4 (No Change) to 7 (Very Much Worse).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (2):
  - AutoCruitment, Atlanta, Georgia
  - Houston Methodist Research Institute, Houston, Texas
- United Kingdom (2):
  - Cambridge University Hospital, Cambridge
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc84db2bf003ab46046